CLINICAL TRIAL: NCT05314166
Title: Impact of Face-to-face Meditation on Non-attachment to Self and Identity Threat
Acronym: MEDIT-PRESENT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2022-RIPH_004_MEDIT-ENPRESENT
Record Dates: First submitted 2022-03-28; First posted 2022-04-06 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Meditation
Keywords: non-attachment to the self; identity threat; face-to-face meditation; focused attention; contemplation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "focused attention" group (Experimental): "focused attention" group: adult subjects practicing face-to-face focused attention meditation.
  Interventions: Other: meditation practice
- "contemplation" group (Active Comparator): "contemplation" group: adult subjects practicing face-to-face contemplation meditation.
  Interventions: Other: meditation practice

INTERVENTIONS:
Other: meditation practice — Description: meditation practice

SUMMARY:
Meditation is widely recognized for its benefits on both physical and psychological health and more particularly on the prevention of depression relapse. However, despite a lot of literature showing its efficacy, the mechanisms of action underlying its benefits have yet to be specifically identified and empirically tested.

to understand these mechanisms actions, it is essential to distinguish meditative practices. Three different categories of meditation can be distinguished: "Attention Family", "Constructive Family" and "Deconstructive Family" with specific effects for each.

DETAILED DESCRIPTION:
The aim of the study is to compare the effects of two types of meditation (focused attention and contemplation) on non-attachment to the self and identity threat

ELIGIBILITY:
Inclusion Criteria:

* male or female
* aged of 18 and more
* without diagnosed psychiatric pathology
* not practicing meditation
* agreeing to participate in the study

Exclusion Criteria:

- less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-05-15 (Estimated); Primary Completion 2023-05-15 (Estimated); Study Completion 2023-07-15 (Estimated)

PRIMARY OUTCOMES:
non-attachment to the self | week 6
  Non-attachment to the self evaluated using Adult Self-transcendence Inventory (ASTI).
  ASTI is composed of 10 items. Each item is coded from 1 (totally disagree) to 7 (totally agree) by comparing how they see life at the time of the questionnaire compared to the last 5 years. The overall score ranges from 10 to 70 points.

SECONDARY OUTCOMES:
Identity threat | week 6
  Identity threat evaluated using Cognitive Appraisal Scale (ECP). ECP is composed of 10 items. Each item is coded from 1 (totally disagree) to 6 (totally agree). The overall score ranges from 6 to 60 points

IPD SHARING:
Plan to Share IPD: No